CLINICAL TRIAL: NCT06927726
Title: Assessment of Anesthetic Efficacy and Hemodynamic Stability of 4% Articaine (1:100,000 Epinephrine) Versus 3% Mepivacaine Used in Maxillary Teeth Extraction for Hypertensive Patients: A Double-blind Randomized Clinical Study
Brief Title: Assessment of Anesthetic Efficacy and Hemodynamic Stability of Two LA Drugs for Hypertensive Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Marwa Taha Ibrahim, Assistant Professor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-2025
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-04

CONDITIONS: Hypertension
Keywords: hemodynamic stability; hypertensive patients; local anesthetic drugs
MeSH Terms: conditions — Hypertension | interventions — Carticaine; Epinephrine; Mepivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4% articaine (1:100,000 epinephrine) (Active Comparator): Local maxillary infiltration anesthesia adjacent to the tooth with extraction will be the anesthetic method used throughout by a vestibular (1.5 ml) and a palatal injection (0.3 ml). The following agents will be applied for anesthetization: Septanest 4% Articaine HCL With 1:100,000 Epinephrine The injections and the extractions will be performed by certified dentists of Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Tanta University.
  Dental extraction will be performed after full anesthesia, tested with a probe on the buccal mucosa, palatal mucosa, and the tooth itself each minute after injection, and after subjective symptoms of numbness by the patient.
  Interventions: Drug: 4% Articaine HCL With 1:100,000 Epinephrine
- 3% mepivacaine (Active Comparator): Local maxillary infiltration anesthesia adjacent to the tooth with extraction will be the anesthetic method used throughout by a vestibular (1.5 ml) and a palatal injection (0.3 ml). The following agents will be applied for anesthetization: Scandonest 3% plain mepivacaine HCL (Septodont, Manufactured By Novocol Pharmaceuticals of Canada). The injections and the extractions will be performed by certified dentists of Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Tanta University.
  Dental extraction will be performed after full anesthesia, tested with a probe on the buccal mucosa, palatal mucosa, and the tooth itself each minute after injection, and after subjective symptoms of numbness by the patient.
  Interventions: Drug: 3% plain mepivacaine HCL

INTERVENTIONS:
Drug: 4% Articaine HCL With 1:100,000 Epinephrine — Preoperative clinically and radiographic examination will be performed for each patient. Local maxillary infiltration anesthesia adjacent to the tooth with extraction will be the anesthetic method used throughout by a vestibular (1.5 ml) and a palatal injection (0.3 ml). The following agents will be applied for anesthetization: Septanest 4% Articaine HCL With 1:100,000 Epinephrine. The injections and the extractions will be performed by certified dentists of Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Tanta University.
  Dental extraction will be performed after full anesthesia, tested with a probe on the buccal mucosa, palatal mucosa, and the tooth itself each minute after injection, and after subjective symptoms of numbness by the patient.
  Other Names: Septanest
  Arms: 4% articaine (1:100,000 epinephrine)
Drug: 3% plain mepivacaine HCL — Preoperative clinically and radiographic examination will be performed for each patient. Local maxillary infiltration anesthesia adjacent to the tooth with extraction will be the anesthetic method used throughout by a vestibular (1.5 ml) and a palatal injection (0.3 ml). The following agents will be applied for anesthetization: Scandonest 3% plain mepivacaine HCL (Septodont, Manufactured By Novocol Pharmaceuticals of Canada). The injections and the extractions will be performed by certified dentists of Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Tanta University.
  Dental extraction will be performed after full anesthesia, tested with a probe on the buccal mucosa, palatal mucosa, and the tooth itself each minute after injection, and after subjective symptoms of numbness by the patient.
  Other Names: Scandonest
  Arms: 3% mepivacaine

SUMMARY:
Pain control in dentistry is an important factor for reducing the fear and anxiety associated with dental procedures. For tooth extraction, it is mandatory to use resources to manage pain and discomfort such as adequate anesthetic techniques . Patient's systemic health conditions and type of local anesthetic drug used, in addition to duration and extension of the extraction procedure are factors which can influence the management of pain in tooth extractions .

Tooth extractions can cause morbidity and changes in hemodynamic parameters to the patient; therefore, it is paramount to carefully select a local anesthetic drug to minimize adverse events . There are a variety of local anesthetics drugs which can meet the specific requirements of different clinical procedures, among them 4% articaine chloridrate with epinephrine at a ratio of 1:100,000. and with and 3% mepivacaine chloridrate without epinephrine, which are largely used in the dental practice and whose clinical safety has already been tested and proved elsewhere

DETAILED DESCRIPTION:
The aim of this prospective study is to compare the anesthetic efficacy and hemodynamic parameters of 4% articaine chloridrate with epinephrine (1:100,000) versus 3% mepivacaine chloridrate without epinephrine in maxillary infiltration for teeth extraction of in controlled hypertensive patients.

Material and Methods The main inclusion criteria for this prospective, randomized, double-blinded clinical study will be patients in need of single tooth extraction owing to caries and/or periodontitis in the maxilla. with controlled hypertension with blood pressure not exceeding values of 160/100 mm Hg. The exclusion criteria will be patients with systemic health problems (e.g uncontrolled hypertension, unstable angina pectoris, recent myocardial infarct (6 months), refractory dysrhythmias, untreated or uncontrolled congestive heart failure), uncontrolled diabetes mellitus, history of allergic reactions to anesthetics drugs, Pregnancy or breastfeeding, and Patients requiring open surgical extractions or with infected teeth were excluded from the study Patients will be selected from Oral and Maxillofacial Surgery Department, Faculty of Dentistry. Tanta University. Equal randomization was achieved with the use of a computer-generated random number list, and signed inform consent will be obtained from every patient included in the study.

Power calculation A study with sixty subjects is reported to have 90% power to detect a difference in success rate of 21% in a continuous outcome measure assuming a significance level of 5% and a correlation of 0.5 between responses from the same subject.

Anaesthetic administration Preoperative clinically and radiographic examination will be performed for each patient. Local maxillary infiltration anesthesia adjacent to the tooth with extraction will be the anesthetic method used throughout by a vestibular (1.5 ml) and a palatal injection (0.3 ml). The following agents will be applied for anesthetization: Septanest 4% Articaine HCL With 1:100,000 Epinephrine and Scandonest 3% plain mepivacaine HCL (Septodont, Manufactured By Novocol Pharmaceuticals of Canada). The injections and the extractions will be performed by certified dentists of Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Tanta University.

Dental extraction will be performed after full anesthesia, tested with a probe on the buccal mucosa, palatal mucosa, and the tooth itself each minute after injection, and after subjective symptoms of numbness by the patient.

Outcome measures of anesthetic success Successful pulp anesthesia is considered to have occurred when no response is obtained to the maximum stimulation (64 reading) of the electric pulp tester during the test period. If a patient declared full numbness (i.e., soft tissue anesthesia), the onset will be subsequently tested. The time taken to reach complete anesthesia will be evaluated with a stopwatch. Treatment will be regarded as being successfully completed when it is associated with no pain. After treatment, the subjective efficiency of anesthesia by means of pain while injecting and pain during treatment to be rated by Heft-Parker visual analog scale (VAS) from 0 (no pain) to 10 (worst pain).

The patient's hemodynamic parameters will be measured by using an automated sphygmomanometer as follows: systolic (SBP) and diastolic blood pressure, Oxygen blood saturation (SO2) , and heart rate (HR) rate pressure product ( before each injection (reading 1), before starting the intervention, i.e. 5 min after the injection (reading 2), and at 10-min intervals (readings 3 and 4).

ELIGIBILITY:
Inclusion Criteria:

* patients in need of single tooth extraction owing to caries and/or periodontitis in the maxilla, with controlled hypertension with blood pressure not exceeding values of 160/100 mm Hg

Exclusion Criteria:

* patients with systemic health problems (e.g uncontrolled hypertension, unstable angina pectoris
* recent myocardial infarct (6 months)
* refractory dysrhythmias
* untreated or uncontrolled congestive heart failure)
* uncontrolled diabetes mellitus
* history of allergic reactions to anesthetics drugs
* Pregnancy or breastfeeding
* Patients requiring open surgical extractions or with infected teeth

Max Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale | 1 hour
  0 represent no pain and 10 represenet severe pain
systolic (SBP) and diastolic blood pressure | 1 hour
  normal 120/80
heart rate | 1 hour
  normal 70
oxygen saturation | 1 hour
  normal 95-98

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of dentistry, Tanta university, Tanta, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No